CLINICAL TRIAL: NCT01961518
Title: Screening an Orthopedic Population for Mildly-affected Individuals With Morquio Syndrome Type A and Maroteaux-Lamy Syndrome
Brief Title: Screening an Orthopedic Population for Mildly-affected Individuals With Morquio Syndrome A and Maroteaux-Lamy Syndrome
Status: Completed | Type: Observational
Sponsor: Greenwood Genetic Center (Other)
Collaborators: Shriners Hospitals for Children (Other); BioMarin Pharmaceutical (Industry)
Responsible Party: Principal Investigator, R. Curtis Rogers, Senior Clinical Geneticst, Greenwood Genetic Center
Other Study IDs: GGC001
Record Dates: First submitted 2013-10-08; First posted 2013-10-11 (Estimated); Last update posted 2015-08-13 (Estimated); Status verified 2015-08

CONDITIONS: Morquio Syndrome A; Maroteaux Lamy Syndrome; MPS IVA; MPS VI
MeSH Terms: conditions — Mucopolysaccharidosis IV; Mucopolysaccharidosis VI

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Consent will be requested for specimen storage (DNA and urine) to allow use of the specimens for future research related or unrelated to the participant's condition.
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to identify patients with Morquio syndrome type A (MPS IVA) and Maroteaux-Lamy syndrome (MPS VI) who may have been missed or misdiagnosed due to atypical clinical features, a milder course, and/or negative urine screening. We will recruit participants who have certain hip and/or joint problems that could potentially be caused by one of these two genetic conditions through a chart review process conducted at Shriners Hospital for Children in Greenville, SC. Diagnostic testing will be performed for each participant to determine if he or she is affected by one of these two conditions. Results will be disclosed to all participants and their legal guardians, and appropriate follow up will be recommended for those who are found to have abnormal results.

ELIGIBILITY:
Inclusion Criteria:

* Eligible participants must currently receive care in the Shriners Hospitals for Children system, and therefore, will be under 19 years of age.
* Eligible participants must have one of the following diagnoses: bilateral Legg-Calve-Perthes disease, bilateral hip dysplasia, multiple joint pain, unidentified skeletal dysplasia
* Eligible participants (or legal guardian) must be able and willing to sign informed consent/assent in English or Spanish.

Exclusion Criteria:

* Participants with one or more or the above inclusion diagnoses who have a specific etiologic diagnosis will not be eligible to participate in this study.
* If we are unable to obtain the necessary specimens, the participant will be removed from the study.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: We plan to recruit 75 patients who will meet chart review criteria, selected from a population of 250-300 patients in the Shriners Hospitals for Children--Greenville (SHC) database. In addition, any patients evaluated at a monthly Genetics clinic held at SHC who meet eligibility criteria will be offered enrollment in the study in person (with a goal of 15). Participants of any ethnicity and both genders will be represented in this study. Since participants will be selected from the SHC patient database, as well as Greenwood Genetic Center clinics held at SHC in Greenville, SC, study participant's geographic location will be concentrated in the Southeastern region of the United States.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2013-10; Primary Completion 2014-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Prevalence of MPS IVA and MPS VI in an pediatric orthopedic population | Data will be reviewed at the end of 1 year
  The primary objective of this study is to identify patients with Morquio syndrome type A or Maroteaux-Lamy syndrome who may have been missed or misdiagnosed due to atypical clinical features, a milder course, and/or negative mucopolysaccharidosis urine screening.

SECONDARY OUTCOMES:
DNA and urine collection and storage in a pediatric orthopedic population | Specimen collection will occur within one year, and specimen storage will be indefinite
  The secondary objective of this study is to obtain and keep blood and urine samples for possible future research on Morquio syndrome type A, Maroteaux-Lamy syndrome, or other related or unrelated diseases.

CONTACTS AND LOCATIONS:
Overall Officials: Richard Curtis Rogers, MD, Principal Investigator — Greenwood Genetic Center
Locations (1):
- Greenwood Genetic Center, Greenville, South Carolina, United States